CLINICAL TRIAL: NCT04806490
Title: Establish and Validate Study of Standard Scale for Syndrome Differentiation of Yin Deficiency Syndrome
Brief Title: Standard Scale for Syndrome Differentiation of Yin Deficiency Syndrome
Acronym: SFYDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: China Academy of Chinese Medical Sciences (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Beijing University of Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2018YFC1704401
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Yin Deficiency Syndrome
Keywords: standard scale; syndrome differentiation; Yin Deficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chinese participants with Yin Deficiency Syndrome: The participants with Yin Deficiency syndrome were included in this study. Chinese Medicine Experts evaluated the main symptoms of Yin Deficiency syndrome, diagnosed those participants.
  And the participants were measured by the standard scale for syndrome differentiation of Yin Deficiency syndrome. The participants were followed up for 12 months to observe whether there were any manifestations of Yin Deficiency syndrome during the observation period.
  Interventions: Diagnostic Test: the diagnosis for Yin Deficiency Syndrome
- Chinese participants without Yin Deficiency Syndrome: The participants without Yin Deficiency syndrome were included in this study. Chinese Medicine Experts evaluated the main symptoms of Yin Deficiency syndrome, diagnosed those participants.
  And the participants were measured by the standard scale for syndrome differentiation of Yin Deficiency syndrome. The participants were followed up for 12 months to observe whether there were any manifestations of Yin Deficiency syndrome during the observation period.
  Interventions: Diagnostic Test: the diagnosis for Yin Deficiency Syndrome

INTERVENTIONS:
Diagnostic Test: the diagnosis for Yin Deficiency Syndrome — The measurement of the standard scale for syndrome differentiation of Yin Deficiency Syndrome

SUMMARY:
An version of the standard scale for syndrome differentiation of Yin Deficiency Syndrome is not available yet for Chinese medicine.

The aim of this study is to develop and validate the standard scale for syndrome differentiation of Yin Deficiency Syndrome. The study is divided into two steps. The first step is to develop the standard scale for syndrome differentiation of Yin Deficiency Syndrome through expert consultation (Delphi method). The second step is to apply the scale in the participants and find out the diagnostic cut-off value of the scale by comparing it with the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be recruited from the current outpatients' clinic activity of the affiliated hospitals of Beijing University of Chinese Medicine and Nanjing University of Chinese Medicine. Subjects must be able to read and write in Chinese. After obtained informed consent we will ask them to participate to this study.
* All the subjects need to fill in the scale of Yin Deficiency syndrome and be diagnosed by a specialist in traditional Chinese medicine (TCM) to determine whether they have Yin deficiency syndrome. The judgment of TCM experts is the gold standard.

Exclusion Criteria:

* Participates who not meet eligibility criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the subjects were enrolled continuously in the TCM outpatient department. If the informed consent of the researcher is obtained, the scale measurement of the study subjects can be carried out.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the diagnostic cut-off value of scale | 12 months
  find out the diagnostic cut-off value of the standard scale for syndrome differentiation of Yin Deficiency Syndrome.

SECONDARY OUTCOMES:
Accuracy of the Standard Scale for Syndrome Differentiation of Yin Deficiency Syndrome | 12 months
  By comparing the consistency between the scale diagnosis and expert diagnosis, the accuracy of the scale diagnosis of Yin deficiency syndrome was judged.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of this study and the publication of relevant research papers, all the research object data in this study will be made public to anyone, but only after de-identification.